CLINICAL TRIAL: NCT01863173
Title: The Effect of Metoprolol Succinate on the Cardiac Function of Patients With Thalassemia Cardiomyopathy a Double Blind Randomized Study
Brief Title: Effect of Metoprolol on Thalassemia Cardiomyopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91-3502
Record Dates: First submitted 2013-05-18; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: B Thalassemia
Keywords: Thalassemia cardiomyopathy; metoprolol succinate; echocardiography; six minute walk test
MeSH Terms: conditions — beta-Thalassemia | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metoprolol (Active Comparator): patient or intervention group
  Interventions: Drug: metoprolol
- placebo group (Active Comparator): control group
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: metoprolol — using B blocker in patient group
  Arms: metoprolol
Drug: placebo — placebo to control group
  Arms: placebo group

SUMMARY:
effect of B blocker was first evaluated in patient with cardiomyopathy not induced by ischemia and idiopathic which as the most common causes of cardiomyopathy. Effect of BB on Thalassemia cardiomyopathy was evaluated in this study

DETAILED DESCRIPTION:
In this clinical trial, 45 patients with thalassemia cardiomyopathy were randomized to receive either metoprolol (n = 26) or placebo (n = 19). Echocardiography and 6 minute walk test was performed at baseline and repeated after 6 months and the values were compared.

ELIGIBILITY:
Inclusion Criteria:

* documented LVEF < 50% by echocardiography
* B thalassemia
* No decompensated heart failure for at least 4 weeks (hospitalization for CHF, worsening lower extremity edema, worsening dyspnea on exertion, , and orthopnea)
* have no evidence of acute myocarditis and
* hemoglobin level above 7 gr⁄dL.

Exclusion Criteria:

* pulse rate below 60/min
* systolic blood pressure less than 90 mmHg
* evidence of peripheral vascular disease
* major depression, history of asthma, PR interval more than 240 msec, second or third degree AV block
* major medical diseases including diabetes mellitus requiring insulin injection, hypothyroidism, hypoparathyroidism, chronic renal failure (glomerular filtration rate below 30 ml/min), hepatic cirrhosis, hepatitis-B and hepatitis-C, positive tests for human immunodeficiency virus, and other hemoglobinopathies

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
ejection fraction | 6 months
  LV contractility
6 minutes walk test | 6 months
  functional capacity
endsystolic volume | 6 months
  functional capacity

SECONDARY OUTCOMES:
patient compliance | 6 months
  drug complication,

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Background] Atiq M, Bana M, Ahmed US, Bano S, Yousuf M, Fadoo Z, Khurshid M. Cardiac disease in beta-thalassaemia major: Is it reversible? Singapore Med J. 2006 Aug;47(8):693-6. PMID 16865210
- [Background] Murphy CJ, Oudit GY. Iron-overload cardiomyopathy: pathophysiology, diagnosis, and treatment. J Card Fail. 2010 Nov;16(11):888-900. doi: 10.1016/j.cardfail.2010.05.009. Epub 2010 Jul 3. PMID 21055653
- [Derived] Kojury J, Zolghadrasli A, Karimi M, Babaee Beighi MA, Namazi S. The effect of metoprolol succinate on the cardiac function of patients with thalassaemia cardiomyopathy: a double-blind randomised study. Heart Asia. 2014 Apr 17;6(1):54-8. doi: 10.1136/heartasia-2013-010460. eCollection 2014. PMID 27326168